CLINICAL TRIAL: NCT06083311
Title: A Randomised, Triple-blinded, Placebo-controlled, Parallel Group Pilot Study, to Assess the Effect of Probiotic on Functional Constipation and Gut Microbiology
Brief Title: The Efficacy of a Probiotic for Functional Constipation (FC)
Acronym: SLOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTB2022TN103
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Functional Constipation
Keywords: Probiotic; GI microbiome; Lactobacillus; Bifidobacterium
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple Blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Participants in this arm will receive a daily dose of 3x10^9 Colony Forming Units (CFU) of a live bacterium, corresponding to 1 capsules daily for 28 days
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants in this arm will receive an equivalent placebo for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants in this arm will receive a daily dose of 3x10^9 Colony Forming Units (CFU) of a live bacterium, corresponding to 1 capsules daily for 28 days
  Arms: Probiotic
Dietary Supplement: Placebo — Participants in this arm will receive an equivalent placebo for 28 days
  Arms: Placebo

SUMMARY:
Investigate the effect of a probiotic (live bacteria) in individuals with functional constipation.

DETAILED DESCRIPTION:
This study aims to investigate the safety and efficacy of live bacteria on defecation parameters in individuals with Functional Constipation. The trial will be run in Germany and will recruit adult men and women meeting the ROME-IV criteria for functional constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Males (at least 30% of total number of subjects) and females ≥ 18 years and ≤65 years old
2. Body Mass Index (BMI) 18.5 - 30.0 kg/m2
3. Fulfilment of the Rome IV FC diagnostic criteria at V1 and V2
4. Self-reported average stool frequency of 3 or less bowel movements per week
5. Self-reported average stool consistency of type 1-4 on the Bristol Stool Form Scale
6. Cleveland Clinic Constipation Score > 8 at V1
7. Readiness not to use any treatment/supplementation for complaints related to constipation (e.g. prokinetics, laxatives, enemas) during the study; exception: glycerol suppository and if it provides no benefit, participants are allowed to take oral laxatives (see section 0)
8. Readiness and ability to comply with and perform the procedures requested by the protocol
9. If receiving proton pump inhibitors (PPI), anticipated to continue PPI therapy for the duration of the trial
10. Readiness not to have any change in habitual diet or exercise patterns over the study period
11. Women:

    * If sexually active, commitment to use contraception methods
    * negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1
12. Generally, in the opinion of investigator, healthy individuals (e.g. no heart failure, no malignancy) Participation is based upon written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Clinically relevant (as per investigators judgement) self-reported chronic disease of the gastrointestinal tract (e.g. irritable bowel syndrome, Crohn's disease, ulcerative colitis, celiac disease, diverticulitis, malabsorption disorder), neurological, cardiovascular, endocrine/reproductive, renal, or other chronic diseases likely to affect gut motility
2. Prior abdominal surgery in the past 3 years (except for laparoscopic appendectomy and cholecystectomy and other minor laparoscopic surgeries, as per investigator judgement, that are allowed)
3. Ongoing regular use of products that (in the investigator's opinion) are known to cause constipation or change gastric motility (e.g. iron; opioids; sucralfate; 5-HT3 antagonists (e.g. ondansetron); antacids with magnesium, calcium, or aluminum; anticholinergic agents; calcium supplements; trycyclic antidepressants; systemic steroids)
4. Any subjects with use of PPI within the last 8 weeks prior to Visit 1 (exception: continuous use for ≥ 8 week before Visit 1 is allowed)
5. Post-menopausal women, defined as >12 months after the last menstrual bleeding and not using hormonal contraception
6. Women ≥ 50 years using hormonal contraception
7. ALARM features in the past 3 months prior to study (e.g. fever, unintentional weight loss ≥5 kg, blood in stool, vomiting) and moderate or severe anorectal problems (e.g. rectal bleeding, pelvic organ prolapse, anal fissures)
8. Previously diagnosed lactose intolerance, gluten intolerance, cow's milk allergy and/or soya-allergy
9. Known allergy or hypersensitivity to any ingredients of the investigational product
10. Consumption of biotic supplements (probiotics, prebiotics, synbiotics or post-biotics) within 2 weeks prior to Visit 1 and during the study
11. Regular consumption of fibre supplements and/or laxatives more than 1x a week
12. Use of laxatives within 48 hrs prior to Visit 1
13. Use of antibiotic within 4 weeks prior to Visit 1 and during the study
14. Ongoing alcohol, drug, or medication abuse
15. Participation in other clinical trials within 4 weeks prior to Visit 1 and during the study
16. Planning travel for >1 week during the study duration
17. Anticipated major changes in diet or exercise during the study
18. Pregnant or lactating or planned to become pregnant during the study period
19. Smoking > 5 cigarettes per week
20. An irregular diet, an abnormal sleep cycle, or other lifestyle abnormalities, as per investigator judgement
21. Individuals who, in the opinion of the investigator, are considered to be incompliant clinical attendees or unlikely for any reason to be able to complete the trial as required
22. Clinically relevant deviation of screening laboratory parameters at V1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Difference in change in Cleveland Clinic Constipation score (total) from baseline (V2) to study end (V3) | Baseline (V2), Day 28 (V3)
  Difference in change in Cleveland Clinic Constipation score (CCCS) (total) from baseline (V2) to study end (V3) between verum and placebo groups. Higher scores in the CCCS indicate worse constipation symptoms. (Max score: 30)

SECONDARY OUTCOMES:
Difference in change in Cleveland Clinic Constipation score (total) at 2 week(s) after V2, compared to V2 | Baseline (V2), Day 14
  Difference in change in Cleveland Clinic Constipation score (CCCS) (total) from 2 weeks after V2 to study end (V3) between verum and placebo groups. Higher scores in the CCCS indicate worse constipation symptoms (Max score: 30)
Difference in change in Patient Assessment of Constipation - Quality of Life score (total) from V2 to V3 | Baseline (V2), Day 28 (V3)
  Difference in change in Patient Assessment of Constipation - Quality of Life (PAC-QOL) score (total) from V2 to V3. Higher scores in the PAC-QOL indicate worse constipation symptoms (Max Score: 112)
Difference in change in Patient Assessment of Constipation - Quality of Life score (total) at 2 week(s) after V2, compared to V2 | Baseline (V2), Day 14
  Difference in change in Patient Assessment of Constipation - Quality of Life (PAC-QOL) score (total) from 2 weeks after V2 to V3. Higher scores in the PAC-QOL indicate worse constipation symptoms (Max Score: 112)
Difference in Patient Assessment of Constipation - Quality of Life domain score from V2 to V3 | Baseline (V2), Day 28 (V3)
  Difference in change in Patient Assessment of Constipation - Quality of Life (PAC-QOL) domain scores (total) from V2 to V3. Higher scores in the PAC-QOL domain scores indicate worse constipation symptoms (varying questions in each domain, each question scored 0 - 4 on Likert scale)
Difference in change in Patient Assessment of Constipation - Quality of Life domain scores at 2 week(s) after V2, compared to V2 | Baseline (V2), Day 14
  Difference in change in Patient Assessment of Constipation - Quality of Life (PAC-QOL) domain scores (total) from 2 weeks after V2 to V2. Higher scores in the PAC-QOL domain indicate worse constipation symptoms (varying questions in each domain, each question scored 0 - 4 on Likert scale)
Difference in change in total reflux symptoms score from V2 to V3 | Baseline (V2), Day 28 (V3)
  Difference in (total) reflux questionnaire scores from V2 to V3. Higher scores in the reflux questions indicate worse reflux symptoms. Max score 10.
Difference in change in total reflux symptoms score at 2 weeks after V2, compared to V2 | Baseline (V2), Day 14
  Difference in (total) reflux questionnaire scores from 2 weeks after V2 to V2. Higher scores in the reflux questions indicate worse reflux symptoms. Max score 10.
Difference in change in reflux symptoms sub-scale score (i.e. individual items) from V2 to V3 | Baseline (V2), Day 28 (V3)
  Difference in (subscale) reflux questionnaire scores from V2 to V3. Higher scores in the reflux questions indicate worse reflux symptoms. Each question is a Likert scale ranging from 1-5. Max score is 5.
Difference in change in reflux symptoms sub-scale score (i.e. individual items) at 2 weeks after V2, compared to V2 | Baseline (V2), Day 14
  Difference in (subscale) reflux questionnaire scores from 2 weeks after V2 to V2. Higher scores in the reflux questions indicate worse reflux symptoms. Each question is a Likert scale ranging from 1-5. Max score is 5.
Difference in proportion of stools in different Bristol Stool Form Scale categories (1-2, 3-4, 5-7) at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Proportion of stool in each Bristol Stool Form Scale (BSFS) category at 1, 2, 3 week(s) after V2 and at V3, each compared to V2. BSFS categories range from 1 - 7, with 1 representing hard stool and 7 representing liquid stool.
Difference in change in mean weekly stool frequency at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Difference in change in mean weekly number of bowel movements at 1, 2, 3 week(s) after V2 and at V3, each compared to V2.
Difference in change in mean weekly number of spontaneous bowel movements (without assistance/ medication) at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Difference in change in mean weekly number of spontaneous bowel movements (without assistance/ medication) at 1, 2, 3 week(s) after V2 and at V3, each compared to V2
Difference in change of the weekly degree of straining (VAS) at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Difference in change of the weekly average degree of straining (VAS) at 1, 2, 3 week(s) after V2 and at V3, each compared to V2. Straining calculated on a 5-point Likert Scale, where 1 is no straining and 5 is very severe straining
Difference in change of the weekly defecation/ rectal pain (VAS) at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Difference in change of the weekly average defecation/rectal pain at 1, 2, 3 week(s) after V2 and at V3, each compared to V2. Defecation/Rectal pain calculated on a 5-point Likert Scale, where 1 is no painand 5 is very severe pain
Difference in the weekly self-assessment of complete bowel emptying at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Difference in the weekly average self-assessment of complete bowel emptying at 1, 2, 3 week(s) after V2 and at V3, each compared to V2. Self assessment of complete bowel emptying conducted with a 'yes' or 'no' question
Difference in weekly average use of laxatives at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Difference in weekly average use of laxatives at 1, 2, 3 week(s) after V2 and at V3, each compared to V2
Difference in weekly need for digital assistance at 1, 2, 3 week(s) after V2 and at V3, each compared to V2 | Baseline (V2), Day 7, Day 14, Day 21 and Day 28
  Difference in weekly average need for digital assistance at 1, 2, 3 week(s) after V2 and at V3, each compared to V2
Difference in short chain fatty acids (SCFA) in stool samples collected prior to V2 and prior to V3 | Baseline (V2), Day 28 (V3)
  Difference in short chain fatty acids (SCFA) in stool samples collected prior to V2 and prior to V3.
Difference in findings of microbiome assessment using metagenomics techniques of stool samples collected prior to V2 and prior to V3 | Baseline (V2), Day 28 (V3)
  Difference in findings of microbiome assessment using metagenomics techniques of stool samples collected prior to V2 and prior to V3
Difference in findings of targeted metabolomic analysis of stool samples collected prior to V2 and prior to V3 | Baseline (V2), Day 28 (V3)
  Difference in findings of targeted metabolomic analysis of stool samples collected prior to V2 and prior to V3
Percentage of subjects with matching records of blinded assessment concern-ing the IP type they received (verum, placebo) and the actual IP assignment | Day 28 (V3)
  Percentage of subjects with matching records of blinded assessment concern-ing the IP type they received (verum, placebo) and the actual IP assignment
Assessment of benefit by subject and investigator at V3 (4 point categorical scale) | Day 28 (V3)
  Assessment of benefit by subject and investigator at V3. 4 point scale, where 1 = poor and 4 = very good
Assessment of the number of adverse events between the intervention and placebo | Day 28 (V3)
  Assessment of the number of adverse events between the intervention and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- analyze & realize GmbH, Berlin, Germany